CLINICAL TRIAL: NCT05711927
Title: The Effect of Sleeping Environment on Sleep-Wake Organization in Preterm Infants
Brief Title: Sleep in SNOO Smart Sleeper Bassinet in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Happiest Baby, Inc. (Industry)
Responsible Party: Principal Investigator, Rakesh Sahni, Medical Director of the Neonatal Intensive Care Unit at NewYork-Presbyterian/Morgan Stanley Children's Hospital, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAU2315
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Prematurity; Very Preterm Maturity of Infant
Keywords: sleep; SNOO; bassinet; white noise; rocking; swaddle; intrauterine environment; crying
MeSH Terms: conditions — Premature Birth; Stereotypic Movement Disorder; Crying

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the traditional bassinet condition or the SNOO Smart Sleeper. Depending on the group to which they are assigned, participants will spend six hours total (divided between two time points) under either the traditional bassinet conditions or in the SNOO Smart Sleeper while having a sleep assessment performed.
  The first sleep assessment will occur at 35-36 weeks postmenstrual age, and the second will occur at term-equivalent age (37 weeks or greater). Each sleep assessment will last three hours and will occur between feeds (2:00 p.m. to 5:00 p.m.).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- SNOO group (Experimental): The SNOO Smart Sleeper will be used in accordance with the manufacturer's programming and instructions.
  Interventions: Device: SNOO Smart Sleeper
- Traditional bassinet group (Sham Comparator): The SNOO will remain powered off to mimic the conditions of sleeping in a traditional hospital bassinet.
  Interventions: Device: Traditional bassinet

INTERVENTIONS:
Device: SNOO Smart Sleeper — Infants will be secured in the SNOO Sleep Sack. They will be placed in the center of the SNOO Smart Sleeper. The SNOO will be powered on and will start playing white noise and rocking from side-to-side. The SNOO's movement and sound settings will automatically ramp up and down as needed in response to the infant's sensed level of fussiness or crying per the manufacturer's programming. The "preemie mode" will be enabled, which caps motion at level 2 out of 5.
  Arms: SNOO group
Device: Traditional bassinet — Infants will be swaddled using a standard hospital blanket. They will be placed in the center of the SNOO Smart Sleeper, but the SNOO will be left powered-off. No white noise will be played. No side-to-side rocking motions will occur.
  Arms: Traditional bassinet group

SUMMARY:
The goal of this clinical trial is to compare sleeping in a SNOO Smart Sleeper bassinet (SNOO) with sleeping in traditional bassinet conditions in premature infants. The main questions it aims to answer are:

1. Do preterm infants who sleep in the SNOO have more quiet sleep?
2. Do preterm infants who sleep in the SNOO have improved vital signs?

   * Participants will spend two separate three-hour periods sleeping in either a SNOO (which plays white noise and rocks from side-to-side) or in a SNOO that remains off (does not play white noise and does not move). There will be at least one week separating these sleep assessments.
   * Participants will have their sleep stage and vital signs monitored (heart rate and oxygen levels).
   * Participants will also wear two stickers on their forehead that measure brain oxygen levels (NIRS) and brain waves (EEG).

There is a chance that the infant may experience more restful sleep and improved vital signs during the 2 sleep assessments.

DETAILED DESCRIPTION:
Sleep plays an important role in the brain growth and development of preterm infants. Neonatal sleep is made up of three stages of sleep: quiet sleep, active sleep, and transitional sleep. Poor sleep can be a result of premature birth itself as well as from simply being in the neonatal intensive care unit (NICU) environment. The interruptions that these infants are exposed to include frequent cares, physical exams, lights, and noises.

The investigators are interested in the potential positive effects on sleep of recreating the environment of the womb. The SNOO is a bassinet that uses the combination of a secure swaddle, white noise, and gentle rocking movements to mimic the conditions that infants were exposed to in the uterus before being born. The investigators are interested in studying how recreating this environment of "within the womb" impacts the sleep-wake cycles of premature infants. To do this, the investigators will measure the amount of time that premature infants spent asleep versus awake while in the SNOO through behavior observations, electroencephalogram (brain activity monitoring), and vital signs. The investigators hypothesize that sleeping in the SNOO will increase the amount of time that the premature infants spend in quiet sleep and will improve their vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients at the Morgan Stanley Children's Hospital NICU.
* Singleton gestation.
* Gestational age 28w0d to 36w6d at birth.
* Postmenstrual age greater than 35 weeks at the time of the intervention.
* Weight greater than 1.8 kg and less than 11.3 kg.
* Stable thermoregulation in an open crib.
* Stable respiratory status on room air (no nasal cannula or CPAP).
* Normal head ultrasound (if obtained).

Exclusion Criteria:

* Congenital brain or spinal anomalies.
* Intracranial hemorrhage.
* Severe encephalopathy.
* Known or suspected genetic syndromes that could result in cerebral dysfunction.
* Airway anomalies that could result in sleep-disordered breathing.
* Bleeding diatheses.
* Status post surgery or minor surgical procedures (i.e. inguinal hernia repair, circumcision).
* Fetal opioid exposure.
* Administration of sedating agents over the past 24 hours.
* Ability to independently roll to hands and knees.

Ages: 1 Week to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Sahni, MD, Principal Investigator — Columbia University
Locations (1):
- Morgan Stanley Children's Hospital Neonatal Intensive Care Unit, NewYork Presbyterian, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calciolari G, Montirosso R. The sleep protection in the preterm infants. J Matern Fetal Neonatal Med. 2011 Oct;24 Suppl 1:12-4. doi: 10.3109/14767058.2011.607563. PMID 21942583
- [Background] Santos J, Pearce SE, Stroustrup A. Impact of hospital-based environmental exposures on neurodevelopmental outcomes of preterm infants. Curr Opin Pediatr. 2015 Apr;27(2):254-60. doi: 10.1097/MOP.0000000000000190. PMID 25635585
- [Background] Zhang X, Spear E, Hsu HL, Gennings C, Stroustrup A. NICU-based stress response and preterm infant neurobehavior: exploring the critical windows for exposure. Pediatr Res. 2022 Nov;92(5):1470-1478. doi: 10.1038/s41390-022-01983-3. Epub 2022 Feb 16. PMID 35173301
- [Background] Johnson S, Marlow N. Preterm birth and childhood psychiatric disorders. Pediatr Res. 2011 May;69(5 Pt 2):11R-8R. doi: 10.1203/PDR.0b013e318212faa0. PMID 21289534
- [Background] Smith GC, Gutovich J, Smyser C, Pineda R, Newnham C, Tjoeng TH, Vavasseur C, Wallendorf M, Neil J, Inder T. Neonatal intensive care unit stress is associated with brain development in preterm infants. Ann Neurol. 2011 Oct;70(4):541-9. doi: 10.1002/ana.22545. Epub 2011 Oct 4. PMID 21976396
- [Background] Restin T, Gaspar M, Bassler D, Kurtcuoglu V, Scholkmann F, Haslbeck FB. Newborn Incubators Do Not Protect from High Noise Levels in the Neonatal Intensive Care Unit and Are Relevant Noise Sources by Themselves. Children (Basel). 2021 Aug 16;8(8):704. doi: 10.3390/children8080704. PMID 34438595
- [Background] Spencer JA, Moran DJ, Lee A, Talbert D. White noise and sleep induction. Arch Dis Child. 1990 Jan;65(1):135-7. doi: 10.1136/adc.65.1.135. PMID 2405784
- [Background] Dereymaeker A, Pillay K, Vervisch J, De Vos M, Van Huffel S, Jansen K, Naulaers G. Review of sleep-EEG in preterm and term neonates. Early Hum Dev. 2017 Oct;113:87-103. doi: 10.1016/j.earlhumdev.2017.07.003. Epub 2017 Jul 12. PMID 28711233
- [Background] Weisman O, Magori-Cohen R, Louzoun Y, Eidelman AI, Feldman R. Sleep-wake transitions in premature neonates predict early development. Pediatrics. 2011 Oct;128(4):706-14. doi: 10.1542/peds.2011-0047. Epub 2011 Sep 12. PMID 21911350
- [Background] Barbeau DY, Weiss MD. Sleep Disturbances in Newborns. Children (Basel). 2017 Oct 20;4(10):90. doi: 10.3390/children4100090. PMID 29053622
- [Background] Kuhn P, Zores C, Pebayle T, Hoeft A, Langlet C, Escande B, Astruc D, Dufour A. Infants born very preterm react to variations of the acoustic environment in their incubator from a minimum signal-to-noise ratio threshold of 5 to 10 dBA. Pediatr Res. 2012 Apr;71(4 Pt 1):386-92. doi: 10.1038/pr.2011.76. Epub 2012 Feb 15. PMID 22391640
- [Background] Zores C, Dufour A, Pebayle T, Dahan I, Astruc D, Kuhn P. Observational study found that even small variations in light can wake up very preterm infants in a neonatal intensive care unit. Acta Paediatr. 2018 Jul;107(7):1191-1197. doi: 10.1111/apa.14261. Epub 2018 Feb 27. PMID 29412484
- [Background] Levy J, Hassan F, Plegue MA, Sokoloff MD, Kushwaha JS, Chervin RD, Barks JD, Shellhaas RA. Impact of hands-on care on infant sleep in the neonatal intensive care unit. Pediatr Pulmonol. 2017 Jan;52(1):84-90. doi: 10.1002/ppul.23513. Epub 2016 Jun 30. PMID 27362468

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SNOO Group | Traditional Bassinet Group
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SNOO Group | Traditional Bassinet Group | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Gestational age
  weeks | 32.9 (1.9) | 33.5 (1.4) | 33.1 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 6 | 4 | 10
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 4 | 2 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percent of Quiet Sleep Time During 3-hour Sleep Assessment
Description: Quiet sleep is a marker of sleep maturation and will be measured by the researcher during the 3-hour-long sleep assessments. Quiet sleep defined as eyes closed with predominantly flaccid "rag doll" appearance, body movements limited to startles, and rhythmic jaw jerks lasting 1 to 2 seconds.
Time Frame: At baseline sleep assessment, up to 3 hours
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | SNOO Group | Traditional Bassinet Group
Number analyzed (Participants) | 11 | 9
percent | 26.8 (9.5) | 19.8 (5.1)

2. Secondary Outcome: Change in Heart Rate Variability
Description: Heart rate variability is the fluctuation of beat-to-beat heart rate intervals over time and is a marker of autonomic nervous system maturation.
Time Frame: Up to 3 hours
Reporting Status: Not Posted, anticipated posting 2026-06

3. Secondary Outcome: Change in Cerebral Oxygenation
Description: Cerebral oxygenation is a measure of the oxygen content of brain and will be measured by near-infrared spectroscopy (NIRS).
Time Frame: Up to 3 hours
Reporting Status: Not Posted, anticipated posting 2026-06

4. Secondary Outcome: Change in Oxygen Saturation
Description: Oxygen saturation is a measure of the oxygen content of the blood, as measured by pulse oximetry.
Time Frame: Up to 3 hours
Reporting Status: Not Posted, anticipated posting 2026-06

5. Secondary Outcome: Change in Intermittent Hypoxemic Event Frequency
Description: Intermittent hypoxemic events are episodes where oxygen saturation is low for prolonged periods, as measured by pulse oximetry.
Time Frame: Up to 3 hours
Reporting Status: Not Posted, anticipated posting 2026-06

ADVERSE EVENTS:
Time Frame: During sleep time (approx 3 hours) at baseline sleep assessment
Arm/Group | SNOO Group | Traditional Bassinet Group
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

LIMITATIONS AND CAVEATS:
All infants were discharged from the NICU after the 1st sleep assessment and were therefore not able to do a 2nd sleep assessment as outlined in the protocol, so the results presented in this record only reflects data collected from one 3-hour sleep assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT05711927/Prot_SAP_000.pdf